CLINICAL TRIAL: NCT05819463
Title: Treatment and Medical Care of Patients With Moderate-to-severe Atopic Dermatitis - Swiss National Clinical Registry TREATswitzerland
Brief Title: Treatment and Medical Care of Patients With Moderate-to-severe Atopic Dermatitis - TREATswitzerland
Status: Recruiting | Type: Observational
Sponsor: Swiss Society of Dermatology and Venereology (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-00205
Record Dates: First submitted 2023-01-23; First posted 2023-04-19 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
As structured and detailed data on the management of AD, a common chronic inflammatory skin disease which has a high impact on patients' quality of life and socioeconomic burden, are not available in Switzerland, the planned registry will overcome this gap. It will provide data on the medical care of patients with AD for health care research and allow to study the efficacy and safety of approved and available therapies for AD in daily life.

DETAILED DESCRIPTION:
A prospective, non-interventional, national multicenter study in patients with moderate-to-severe AD. According to the availability of approved systemic drugs for the treatment of AD, the study will include children ≥12 years, adolescents and adult patients.

The general goal of the AD registry TREATswitzerland is to provide the scientific community with a disease-oriented prospective cohort of patients suffering from moderate-to-severe AD.

The primary objective of the AD registry is the documentation of medical care given to patients with moderate-to-severe AD in order to assess the appropriateness of care.

Further objectives of the AD registry are:

1. to evaluate the psychosocial impact of AD;
2. to provide up-to-date epidemiologic data that allow investigating risk factors for favorable or unfavorable disease courses and comorbidities; and
3. to establish a research network and foster clinical research projects.

The study procedures include:

* No study related intervention will be performed
* Patients have to fulfill all inclusion criteria to be enrolled in the study.
* Included patients are prospectively followed for at least 24 months. A maximum duration of follow-up is not intended.
* During the observation period, standardized study visits are performed to prospectively document patient characteristics, clinical data, patient-reported outcomes, reasons for treatment decisions, and satisfaction with treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 12 years
* AD according to the UK Working Party's Diagnostic Criteria (28)
* Moderate to severe AD as defined by
* objective SCORAD > 20 or IGA ≥ 3 (moderate) or
* currently on systemic antiinflammatory therapy for AD or
* previous systemic antiinflammatory therapy for AD within past 24 months

Exclusion Criteria:

* refusal to sign the informed consent form

Min Age: 12 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The study aims at including 700 patients with moderate to severe atopic dermatitis in the registry.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2022-06-02 (Actual); Primary Completion 2032-05 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the type of systemic therapy used in patients with moderate-to-severe atopic dermatitis | 24 months
  assess medical substances given systemically to treat AD

SECONDARY OUTCOMES:
assessment of patients demographic data | 24 months
  assess sex (male, female), age (years)
assessment of past treatment and current treatment | 24 months
  assess specific medical substances (name, dosage, duration of therapy, clinical effects, adverse effects)
assessment of concomitant topical therapy for AD and concomitant treatment | 24 months
  describe medical substances given for AD skin therapy (e.g. topical corticosteroids) and topical calcineurin inhibitors), and medical substances given for concomitant diseases
assessment of past and current comorbidities | 24 months
  describe diseases
change in subjective and objective SCORAD (SCORing Atopic Dermatitis) | 24 months
  outcome measure for disease severity
change in EASI (Eczema Area and Severity Index) | 24 months
  Investigator-assessed outcome measure for disease severity
change in DLQI (Dermatology Life Quality Index) | 24 months
  Patient-reported outcome measure for skin-related quality of life
change in POEM (Patient Oriented Eczema Measure) | 24 months
  Patient-reported outcome measure for atopic eczema severity
change in RECAP (Recap of atopic eczema) | 24 months
  Patient-reported outcome measure to capture eczema control

CONTACTS AND LOCATIONS:
Overall Officials: Dagmar Simon, Prof. Dr. med., Principal Investigator — Department of Dermatology, Inselspital
Locations (9):
- Switzerland (9):
  - Universitätsspital Basel, Allergologie, Basel
  - Inselspital, Department of Dermatology, Bern
  - Dermatology & Skin Care Clinic, Buochs
  - HFR Hôpital Cantonal de Fribourg, Fribourg
  - Dermatologie CHUV, Lausanne
  - Luzerner Kantonsspital, Zentrum für Dermatologie und Allergologie, Lucerne
  - Kantonsspital St. Gallen - Klinik für Dermatologie, Venerologie und Allergologie, Sankt Gallen
  - PLAZA Kliniken, Uster
  - Institut für Dermatologie und Venerologie Stadtspital Zürich Europaallee, Zurich